CLINICAL TRIAL: NCT06645639
Title: Towards Implementation of the Pediatric Integrated Nutrition Pathway for Acute Care Pathway (P-INPAC) - Pilot Study
Brief Title: Implementation of P-INPAC
Acronym: P-INPAC
Status: Recruiting | Type: Observational
Sponsor: The Hospital for Sick Children (Other)
Collaborators: McMaster Children's Hospital (Other); St. Justine's Hospital (Other)
Responsible Party: Principal Investigator, Jessie Hulst, Staff Physician, The Hospital for Sick Children
Other Study IDs: 1000079853
Record Dates: First submitted 2024-07-24; First posted 2024-10-17 (Actual); Last update posted 2024-10-17 (Actual); Status verified 2024-07

CONDITIONS: Malnutrition, Child; Nutrition Poor
MeSH Terms: conditions — Child Nutrition Disorders; Malnutrition

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (3):
- Audit Group: We will perform an audit of health records of all hospitalized patients at one selected study ward, one day of every other week, at each of the 3 study sites to track their routine nutrition care in phase 1 and changes in nutrition care post-implementation in phase 3.
  Interventions: Other: Pediatric Integrated Nutrition Pathway for Acute Care Pathway (P-INPAC)
- Detailed Patient Group: Patients will be recruited in this group from one selected study ward, one day of every other week, at each of the 3 study sites to track their routine nutrition care in phase 1 and changes in nutrition care post-implementation in phase 3. They will also be followed up over a phone call one month after discharge.
  Interventions: Other: Pediatric Integrated Nutrition Pathway for Acute Care Pathway (P-INPAC)
- Healthcare Provider Group: A questionnaire assessing the knowledge, attitude, and self-perceived practices (KAP) amongst healthcare professionals will be conducted with staff, including trainees, at each site's study ward. Further, the workload of the study ward's Registered Dietitian will be assessed for 3 days.

INTERVENTIONS:
Other: Pediatric Integrated Nutrition Pathway for Acute Care Pathway (P-INPAC) — The pediatric working group of Canadian Malnutrition Task Force has developed an evidence-informed algorithm named the Pediatric Integrated Nutrition Pathway for Acute Care (P-INPAC). The P-INPAC outlines a process to improve nutrition care by:
  1. implementing nutrition screening at point-of-admission
  2. introducing standard care measures to prevent the development of malnutrition in children admitted with normal nutrition status, including standardizing the process of monitoring food intake early and systematically to identify when standard care measures are not sufficient
  3. ensuring the moderately and severely malnourished patients receive timely specialized care in the form of a comprehensive assessment and treatment; and
  4. ensuring moderately and severely malnourished patients receive adequate post discharge follow-up and nutrition care.
  In this pilot study, we will be implementing the first two steps of P-INPAC only (screening and assessment).
  Groups: Audit Group; Detailed Patient Group

SUMMARY:
The framework for Pediatric Integrated Nutrition Pathway for Acute Care (P-INPAC) was developed by the Canadian Malnutrition Task Force (CMTF); however, it has not been implemented in a research setting. The framework by CMTF for Integrated Nutrition Pathway for Acute Care (INPAC) in adults was also implemented in the "More-2-Eat" project which led to development of best practices in nutritional culture of the hospitals. Therefore, we intend to undertake this feasibility project at 3-sites to train staff and evaluate the implementation of P-INPAC components as part of routine healthcare procedure.

DETAILED DESCRIPTION:
The P-INPAC pilot study will be a 3-phase multi-center research study in hospitalized children, conducted at The Hospital for Sick Children, Toronto, and two other Canadian pediatric centres: Centre hospitalier universitaire Sainte-Justine, Montreal, Quebec and McMaster Children's Hospital, Hamilton, Ontario. P-INPAC is an algorithm which helps to identify, assess, and treat children with malnutrition.

In the first phase of the study, we will perform an audit of health records of all hospitalized patients at one selected study ward, one day of every other week for 8 weeks, at each of the 3 study sites to track their routine nutrition care. We anticipate auditing 80-100 patients/site in this cycle (total 240-300 patients). In addition, ≈12- 20 patients/ site (≈ 60 in total) who consent to detailed malnutrition screening and assessment would also be identified, assessed, and followed up one month after discharge. In addition, a questionnaire assessing the malnutrition knowledge, attitude, and self-perceived practices (KAP) amongst healthcare professionals will be conducted with staff, including trainees, at each site's study ward. Further, the workload of the study ward's Registered Dietitian (RD) will be assessed for 3 days.

In the second phase of the study, the health care team from each site's study ward will be trained by the site implementation research team about the P-INPAC, and how to administer nutritional screening and perform nutritional assessments, which is the Subjective Global Nutrition Assessment (SGNA).

Finally, in the third phase, we will monitor and evaluate the implementation of the first 2 steps of the P-INPAC (screening & assessment) over a period of 4 months assessing the acceptability, adoption, and coverage of improved nutrition care practices on the same pediatric study wards. We anticipate auditing 160-200 patients/site in this cycle (total 480-600 patients). In addition, detailed patient level data collection will take place in a selected group of consented patients, ≈24-40 patients per site from the 3 sites (≈120 in total). We would also follow-up with these patients a month after discharge.

Healthcare providers will be invited to answer the KAP questionnaire post-implementation version. We will compare responses from phase 1 with phase 3 (pre-/ post-follow up). And, the workload of the ward RD will be assessed again over 3 days.

ELIGIBILITY:
Phase 1 and Phase 3 - Audited patient group inclusion Criteria:

1. ≥ 30 days of age and less than18 years of age on day of assessment
2. Anticipated Length of hospital stay ≥24 hours from day of assessment

Phase 1 & Phase 3 Detailed patient group inclusion Criteria:

1. Admitted to either a general medical or surgical ward
2. ≥ 30 days of age and less than 18 years of age on day of assessment
3. Anticipated Length of stay ≥ 24 hours from day of assessment
4. Speak English (or French at Quebec site) or have a family proxy available at the meal to provide information if first language of patient is not English (or French at Quebec site)
5. Patient/ caregiver provides written consent to participate

Exclusion Criteria:

a. Patients with eating disorder, somatization disorders, ARFID, FORM 1 etc. where the study interaction might interfere with the messaging or therapeutic plan as set out by the responsible team.

Phase 1 and 3 for Health Care Providers inclusion criteria:

1. Implied consent to participate by completing the KAP questionnaire
2. Providing clinical service for the select ward

Ages: 30 Days to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: 2 Patient Groups (Audit and Detailed)
  1 Health care providers group comprising of all the healthcare providers on the participating wards.
Sampling Method: Non-Probability Sample
Enrollment: 600 (Estimated)
Dates: Start 2023-09-04 (Actual); Primary Completion 2025-02-28 (Estimated); Study Completion 2025-12-01 (Estimated)

PRIMARY OUTCOMES:
Baseline nutrition risk screening using STRONGkids or PNST | 2-month period (phase 1)
  Determine routine standard nutritional care practices related to nutrition risk screening in hospitalized children during phase 1 of study using a validated tool, such as, STRONGkids or PNST.
Baseline nutrition risk screening using weight | 2-month period (phase 1)
  Determine routine standard nutritional care practices related to nutrition risk screening in hospitalized children during phase 1 of study using routine anthropometrics - weight
Baseline nutrition risk screening using height or length | 2-month period (phase 1)
  Determine routine standard nutritional care practices related to nutrition risk screening in hospitalized children during phase 1 of study using routine anthropometrics - height or length in children under 2 years of age
Baseline nutrition risk screening using head circumference | 2-month period (phase 1)
  Determine routine standard nutritional care practices related to nutrition risk screening in hospitalized children during phase 1 of study using routine anthropometrics - head circumference in children under 2 years of age
Determine baseline knowledge among healthcare providers using the KAP questionnaire | 2-month period (phase 1)
  Determine baseline knowledge among healthcare providers on recognizing malnutrition and its management in hospitalized children, including perceived barriers and practices, using the KAP questionnaire
Determine changes in knowledge among healthcare providers using the KAP questionnaire | 4-month period (phase 3)
  Determine changes in knowledge among healthcare providers on recognizing malnutrition and its management in hospitalized children in Phase 3, including perceived barriers and practices, using the KAP questionnaire after training was completed in phase 2
Determine success with training and feasibility of nutrition risk screening in hospitalized children using STRONGkids and PNST | 4-month period (phase 3)
  Determine success with training and feasibility of implementing the P-INPAC framework by assessing changes in standard nutritional care practices related to nutrition risk screening in hospitalized children during phase 3 of study using a validated tool, such as, STRONGkids and PNST
Determine success with training and feasibility of nutrition risk screening in hospitalized children using weight | 4-month period (phase 3)
  Determine success with training and feasibility of implementing the P-INPAC framework by assessing changes in standard nutritional care practices related to nutrition risk screening in hospitalized children during phase 3 of study using routine anthropometrics - weight
Determine success with training and feasibility of nutrition risk screening in hospitalized children using height/ length | 4-month period (phase 3)
  Determine success with training and feasibility of implementing the P-INPAC framework by assessing changes in standard nutritional care practices related to nutrition risk screening in hospitalized children during phase 3 of study using routine anthropometrics - height or length in children under 2 years of age
Determine success with training and feasibility of nutrition risk screening in hospitalized children using head circumference | 4-month period (phase 3)
  Determine success with training and feasibility of implementing the P-INPAC framework by assessing changes in standard nutritional care practices related to nutrition risk screening in hospitalized children during phase 3 of study using routine anthropometrics - head circumference in children under 2 years of age

CONTACTS AND LOCATIONS:
Locations (3):
- Canada (3):
  - McMaster Children's Hospital, Hamilton, Ontario
  - The Hospital for Sick Children, Toronto, Ontario
  - Ste-Justine UHC, Montreal, Quebec

IPD SHARING:
Plan to Share IPD: Yes
The data entered the REDCap data collection form will be completely confidential and de-identified and can only be rendered identifiable by linking the study IDs in the data collection form to the study IDs encrypted master linking log. The master linking log will be maintained by the site and not shared by the other site. Confidentiality will be respected and no information that discloses the identity of the participants will be released or published. The data will be kept stored for a minimum of 7 years following collection of the study in accordance with SickKids data retention policy, or longer as per study site institutional research ethics board requirements.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: The data will be kept stored for a minimum of 7 years following collection of the study in accordance with SickKids data retention policy, or longer as per study site institutional research ethics board requirements.
Access Criteria: Research team members

REFERENCES:
- [Background] Hulst JM, Zwart H, Hop WC, Joosten KF. Dutch national survey to test the STRONGkids nutritional risk screening tool in hospitalized children. Clin Nutr. 2010 Feb;29(1):106-11. doi: 10.1016/j.clnu.2009.07.006. Epub 2009 Aug 13. PMID 19682776
- [Background] Secker DJ, Jeejeebhoy KN. How to perform Subjective Global Nutritional assessment in children. J Acad Nutr Diet. 2012 Mar;112(3):424-431.e6. doi: 10.1016/j.jada.2011.08.039. Epub 2012 Mar 1. PMID 22717202
- [Background] Huysentruyt K, Brunet-Wood K, Bandsma R, Gramlich L, Fleming-Carroll B, Hotson B, Byers R, Lovelace H, Persad R, Kalnins D, Martinez A, Marchand V, Vachon M, Hulst JM, On Behalf Of The Canadian Malnutrition Task Force-Pediatric Working Group. Canadian Nationwide Survey on Pediatric Malnutrition Management in Tertiary Hospitals. Nutrients. 2021 Jul 30;13(8):2635. doi: 10.3390/nu13082635. PMID 34444796
- [Background] Keller H, Laur C, Atkins M, Bernier P, Butterworth D, Davidson B, Hotson B, Nasser R, Laporte M, Marcell C, Ray S, Bell J. Update on the Integrated Nutrition Pathway for Acute Care (INPAC): post implementation tailoring and toolkit to support practice improvements. Nutr J. 2018 Jan 5;17(1):2. doi: 10.1186/s12937-017-0310-1. PMID 29304866
- See also: P-INPAC Pathway — https://nutritioncareincanada.ca/resources-and-tools/pediatrics/p-inpac/pathway